CLINICAL TRIAL: NCT02015247
Title: Functional Capacity After Computer Assisted Periacetabular Osteotomy in Patients With Hip Dysplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Functional capacity PAO
Record Dates: First submitted 2013-07-09; First posted 2013-12-19 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2013-08

CONDITIONS: Hip Dysplasia
MeSH Terms: conditions — Hip Dislocation | interventions — Surgery, Computer-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- computer-assisted surgery (Other): use of computer-assisted navigation during periacetabular osteotomy
  Interventions: Procedure: computer-assisted surgery

INTERVENTIONS:
Procedure: computer-assisted surgery — use of computer-assisted navigation during periacetabular osteotomy

SUMMARY:
Pathogenesis of hip dysplasia Hip dysplasia is multifactorial in origin influenced by genetic and intrauterine factors, such as mechanical (rump presentation and oligohydramnios) and hormonal factors1. To ease the passage through the birth canal, the hip joint is quite mobile perinatally. Postnatally, the laxity of the ligaments will subside and the femoral head will normally position itself deeply in the acetabulum2. The theory is that if the femoral head does not migrate sufficiently into the acetabulum, dysplasia may develop because the matrice to stimulate acetabular growth is not correctly positioned. Normally, at birth the femoral head sits deep in the acetabulum held by surface tension of the synovial liquid. The growth and the hemispherical morphology of acetabulum are dependent on the presence of a normally growing and correctly placed spherical femoral head that works as a convex matrice. If for some reason the normal development is disturbed pre- or postnatally, pathologic relations may develop between the femoral head and the acetabulum3, leading to hip dysplasia.

Purpose of this research project is to investigate if the correction of the acetabulum is accurately performed when the surgeon use navigation equipment during PAO.

DETAILED DESCRIPTION:
Morphological changes in hip dysplasia The dysplastic hip joint has a complex morphology characterised by a wide shallow acetabular cavity with an excessively oblique articulating roof. The acetabular cover of the femoral head is globally deficient4;5 and the acetabular rim is hypertrophied possibly due to excessive pull from the often hypertrophic labrum. Anteversion is normal5-7, but occasionally the acetabulum is retroverted8;9. The weight-bearing area between the acetabular roof and head is reduced and the articular cartilage is significantly thicker than normal10. Hip dysplasia is often associated with increased anteversion of the femoral neck5;11 and with valgus neck-shaft angle that results in a reduced abductor lever arm12. However the deformities vary from individual to individual and retroversion of the femoral neck has also been reported in hip dysplasia12. Patients with hip dysplasia are prone to developing osteoarthritis of the hip at a young age 13;14. The reasons for this are not fully understood, but an explanation could be that the reduced contact area between acetabulum and the femoral head as well as a reduced abductor lever arm increase the load per contact-area in the hip joint4. The increased load is a strain on the articular cartilage and believed to result in degeneration of cartilage and the subchondral bone and eventually osteoarthritis14-17. The purpose of periacetabular osteotomy (PAO) is to increase acetabular cover of the femoral head and thereby distribute pressures better over the available cartilage surface.

PAO followed by rehabilitation At PAO, the pubic bone is osteotomized and under fluoroscopic control, the ischial osteotomies and the posterior iliac osteotomy are performed. The acetabular fragment is repositioned to optimise coverage of the femoral head. The repositioning is very challenging and clearly the most demanding aspect of the procedure18. Four weeks after discharge, the rehabilitation is initiated and carried out by two physiotherapists specialised in orthopaedics. The patients come to the hospital for physiotherapy twice a week and each exercise session is 1 hour with a 30-minute aerobic and strength program followed by a 30-minute program of mobility and gait training. Physiotherapy is ended 2-3 months after PAO when the physiotherapists assess that the patient has achieved predetermined functional goals e.g. walking at speed without crutches and ability to run. As a result of the patients' young age, they have had a high physical function and it is the aim, that they will regain this level of function after PAO. It is not yet examined whether PAO patients after surgery attain the functional capacity comparable to the age- and gender-matched population.

ELIGIBILITY:
Inclusion Criteria:

* Radiological diagnosed dysplasia (i.e. centre-edge angle < 25 degrees)
* osteoarthritis degree ≤ 1 according to the criteria of Tonnis
* pain from hip
* minimum 110 degrees flexion in the hip and good rotation
* closed growth zones in the pelvis

Exclusion Criteria:

* neuromuscular diseases
* previously major hip surgery
* pain in the leg (>3 on VAS) other than from the hip
* persons with cognitive problems
* persons unable to speak or understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-12; Primary Completion 2014-11 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
correction of acetabular fragment in 3D | 4 months postop
  position of acetabular fragment measured in three dimensions

SECONDARY OUTCOMES:
functional capacity | 1 year postop
  measured in functional tests with inertia-based measurement analysis

OTHER OUTCOMES:
activity | 4 and 12 months postop
  activity measured with 3-axial accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Søballe, DMSc, Study Director — University of Aarhus; Inger Mechlenburg, PhD, Principal Investigator — University of Aarhus; Inger Mechlenburg, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark